CLINICAL TRIAL: NCT03222882
Title: Transcriptomic Profile of Endometrium in Different Histological Dating of Hormone Replacement Cycle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KYXM-201702-01
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RIF group (Experimental): According to the histological dating and transcriptomic profile of endometrium of hormone replacement cycle in control group, to explore the effectiveness of intervention by advanced or delayed personal embryo transfer . The establishment of standard control group: Frozen embryo transfer patients according to the inclusion and exclusion criteria were evaluated for histological dating and transcriptomic profile by endometrial biopsy on day P＋7 in an HRT cycle. After routine time transfer in the frozen embryo transfer cycle, the standard of histological dating and transcriptomic profile were determined according to the pregnancy outcome of the FET cycle .
  Interventions: Procedure: personal embryo transfer

INTERVENTIONS:
Procedure: personal embryo transfer — According to the histological dating and transcriptomic profile of endometrium of hormone replacement cycle in control group, to explore the effectiveness of intervention by advanced or delayed personal embryo transfer . The establishment of standard control group: Frozen embryo transfer patients according to the inclusion and exclusion criteria were evaluated for histological dating and transcriptomic profile by endometrial biopsy on day P＋7 in an HRT cycle. After routine time transfer in the frozen embryo transfer cycle, the standard of histological dating and transcriptomic profile were determined according to the pregnancy outcome of the FET cycle .

SUMMARY:
At present, the evaluation criterion of endometrial receptivity is controversial. The development of a molecular diagnostic tool, the endometrial receptivity array (ERA) for diagnosis of endometrial receptivity . But use of this test in patients with RIF has shown that the window of implantation (WOI) is displaced in only a quarter of these patients and use of a personalized embryo transfer (pET) on the day designated by ERA improves reproductive performance with higher cost .what is known to the others'population? The morphological changes observed on histology for each specific day after ovulation were described by Noyes and his colleagues in 1950 . An endometrial biopsy that shows a difference of more than 2 days between the histologic dating and actual day after ovulation is considered to be ''out of phase''. But such pET studies according to the Noyes criterion in hormone replacement cycle are lacking . The aim of this study is to explore the transcriptomic profile of endometrial receptivity in different histological dating of hormone replacement cycle and its clinical application.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for RIF group were: unexplained repeated implantation failure (RIF) is defined as the absence of a gestational sac on ultrasound at 5 or more weeks after embryo transfer (ET) after 3 embryo transfers with high quality embryos or after the transfer of ≥10 embryos in multiple transfers.

The inclusion criteria for control group were: (1) age <35 years; (2) unregular menstrual cycles of >37 days; (3) baseline follicle- stimulating hormone (FSH) < 9.0 IU/L; (4) endometrial thickness ≥7.0 mm on the day of hCG administration.

Exclusion Criteria:

* The exclusion criteria were: (1) uterine abnormalities (double uterus, bicornuate uterus, unicornuate uterus); (2) intrauterine adhesions（moderate - severe）, endometriosis, adenomyosis, untreated hydrosalpinx, uterine fibroids (submucosal fibroids, nonmucosal fibroids >4.0 cm and/or endometrial pressure) (3) history of adverse pregnancy (including spontaneous abortion, stillbirth, and fetal malformation).

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 143 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | at least one intrauterine gestational sac with cardiac action by ultrasound performed 28 days after embryo transfer
  clinical pregnancy rate

SECONDARY OUTCOMES:
Biochemical pregnancy | 14 days after embryo transfer
  Biochemical pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: yuan li, Study Chair — Reproductive & Genetic Hospital of CITIC-Xiangya
Locations (1):
- Reproductive & Genetic Hospital of CITIC-XIANGYA, Changsha, Hunan, China